CLINICAL TRIAL: NCT06024915
Title: A Phase I Study to Evaluate Drug-Drug Interaction of TQ05105 Tablets
Brief Title: A Study to Evaluate Drug-Drug Interaction of TQ05105 Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQ05105-I-04
Record Dates: First submitted 2023-08-30; First posted 2023-09-06 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — Itraconazole; Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Itraconazole drug-durg interaction (DDI) (Experimental): Itraconazole capsule: 0.2g once daily on Days 2 to Day 5; TQ05105 tablets: single oral dose on Days 1 and Day 5.
  Interventions: Drug: TQ05105 tablets; Drug: Itraconazole capsule
- Rifampicin DDI (Experimental): Rifampicin Capsule: 0.6g once daily on Days 2 to Day 9; TQ05105 tablets: single oral dose on Days 1 and Day 9.
  Interventions: Drug: TQ05105 tablets; Drug: Rifampicin Capsule

INTERVENTIONS:
Drug: TQ05105 tablets — TQ05105 is a Janus kinase 2 (JAK2) inhibitor.
Drug: Itraconazole capsule — Itraconazole is a strong inhibitor of cytochrome P450 3A (CYP3A).
  Arms: Itraconazole drug-durg interaction (DDI)
Drug: Rifampicin Capsule — Rifampicin is a strong inducer of CYP3A.
  Arms: Rifampicin DDI

SUMMARY:
This is a single-center, open, single-dose, self-controlled phase I clinical trial to evaluate the effects of metabolic enzyme inhibitors/inducers on in vivo metabolic and elimination of TQ05105 tablets, and the safety of metabolic enzyme inhibitors/inducers combined with TQ05105 tablets.

ELIGIBILITY:
Inclusion Criteria:

* At the time of signing the informed consent, males or females between 18 and 45 years of age;
* Female weight ≥ 45 kg, male weight ≥ 50 kg, with a body mass index (BMI) between 19 and 26 kg/m2.
* Subjects in good health, as determined by a medical history, vital signs, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations;
* Subjects can comply with the study procedures, voluntarily participate in the study, and sign the informed consent in person.

Exclusion Criteria:

* Subjects: preexisting or existing circulatory system, endocrine system, nervous system, digestive system, respiratory system, genitourinary system, hematology, immunology, psychiatry and metabolic disorders or abnormalities, or related chronic or acute diseases, the investigator assesses that it is not appropriate to participate in the trial；
* Subjects with Systemic/local acute infection before taking the study drug;
* Subjects who have a history of specific allergies, or allergic conditions (such as allergies to two or more drugs, environments, or foods), or are known to be allergic to components or analogs of the study drug;
* Subjects who have difficulty in swallowing or have any gastrointestinal disorder that affects drug absorption at the time of screening；
* Subjects who cannot receive venous indwelling needle for blood sample collection；
* Subjects who drank regularly in the 6 months prior to first dosing, such as those who drank more than 14 units of alcohol per week or who had a positive alcohol breath test at the time of screening；
* Subjects who had a history of major surgery, or had taken the study drug, or had participated in other drug clinical trials within 3 months prior to initial dosing；
* Subjects who donated blood or lost significant amounts of blood within 3 months prior to initial dosing；
* Subjects who had used drugs within 3 months prior to first dosing, or tested positive for drugs, or had a history of drug abuse within 5 years prior to screening；
* Subjects who smoked more than 5 cigarettes per day in the 3 months prior to initial dosing or who could not stop using any tobacco products during the trial；
* Subjects who consumed excessive amounts of tea, coffee, and/or caffeinated beverages daily in the 30 days prior to initial dosing；
* Subjects who have used any drug that inhibits or induces liver metabolism of the drug in the 30 days prior to initial dosing；
* Subjects who have taken any prescription, over-the-counter, herbal, or health product in the 14 days prior to initial dosing；
* Subjects who have taken a special diet or other factors affecting drug absorption, distribution, metabolism, or excretion within 7 days prior to initial dosing；
* Subjects who ingested chocolate, any caffeinated, or xanthine-rich food or drink 48 hours before first dosing；
* Subjects who have special dietary requirements and cannot follow a uniform diet；
* Female subjects of child-bearing potential；
* Subjects judged by the investigator to be unsuitable to participate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | Up to 10 days.
  Maximum plasma drug concentration after administration.
Time to reach Cmax (Tmax) | Up to 10 days.
  Time to reach the maximum plasma concentration after administration.
Elimination half-life (t1/2) | Up to 6 days.
  The elimination half-life (t1/2) after oral dose of TQ05105 tablets and Itraconazole capsule.

SECONDARY OUTCOMES:
Occurrence of adverse events (AE) | Up to 30 days.
  Including all adverse events (AE) and serious adverse events (SAE).

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China